CLINICAL TRIAL: NCT06295198
Title: Investigation of the Effects of Different Talocrural Mobilization Techniques on Jumping Performance and Kinesiophobia in Professional Basketball Players With Lateral Ankle Sprain -Randomized Single-Blind Study
Brief Title: The Effect of Different Talocrural Joint Mobilization Techniques in Lateral Ankle Sprain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Pelin Pişirici, Assistant Professor, PT, PhD, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OPMM-Ankle Instability
Record Dates: First submitted 2024-02-06; First posted 2024-03-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Ankle Sprains; Ankle Injuries; Kinesiophobia; Jumping From Height
Keywords: talocrural joint; single-leg drop jump test; dorsiflexion limitation
MeSH Terms: conditions — Ankle Injuries; Kinesiophobia

STUDY DESIGN:
Intervention Model Description: Participants with lateral ankle sprains will be randomized to the Mulligan and Maithland groups, and their evaluations and treatments will be completed.
Who Masked: Outcomes Assessor
Masking Description: After evaluations, the groups determined as a result of randomization via a website were placed in opaque envelopes. The participant is randomized to one of the Mulligan or Maitland groups by selecting an envelope.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulligan Group (Experimental): Participants in the Mulligan group stood in front of the physical therapist at the end of the treatment table and placed their affected lower extremity forward and the other slightly backward. The physical therapist placed both hands on top of each other on the patient's talus to stabilize the talus. The athlete was asked to move until he reached the end of his pain-free ankle dorsiflexion range. Meanwhile, the physiotherapist gave posterior pushing with both hands. The Mulligan mobilization technique was performed 10 times by each athlete.
  Interventions: Other: Single lep drop jump test
- Maitland Group (Experimental): Maitland group, III. degree talus mobilization technique was applied. In this mobilization technique, 120 seconds of application, 60 seconds of rest, and then 120 seconds of application were performed. Maitland III, which takes 5 minutes in total. For the 10-degree mobilization technique, the participant was placed on his back with the foot pointing forward, the ankle was placed in 20° plantar flexion, and the talocrural ligament was in a relaxed position. The hand stabilizing the foot was placed proximal to the malleolus to stabilize the leg. The other hand performing the mobilization grasped the anterior talus using the first web space. The talus was then shifted posteriorly downwards with force.
  Interventions: Other: Single lep drop jump test

INTERVENTIONS:
Other: Single lep drop jump test — All evaluations will be repeated before and after the treatment.
  Other Names: Weight-bearing lunge test; Tampa kinesiophobia scale; Fear Avoidance Belief Questionnaire

SUMMARY:
Decreased ankle dorsiflexion range of motion (DFROM) has been identified among the factors that increase the risk of lateral ankle sprain (LAS) in basketball players. Restoring the DFROM is important in restoring reduced functional abilities and reducing the risk of re-injury. There is evidence that talocrural joint mobilization improves DFROM, but studies investigating the effectiveness of different mobilization techniques are needed. Our study aims to investigate the effects of single-session Mulligan and Maitland talocrural joint mobilization methods on dorsiflexion joint range of motion, jumping performance, and kinesiophobia in elite basketball players.

DETAILED DESCRIPTION:
Lateral ankle sprain (LAS) accounts for 80% of all ankle injuries. LAS injuries have high recurrence rates and are the most common injury type in basketball players with a rate of 41.1%. Many LAS injuries; It occurs in situations such as falling to the ground after jumping, at the end of the swing phase, during contact of the foot with the ground, in hard turns, collision, falling and sudden stopping. Decreased ankle dorsiflexion range of motion has been identified among the factors that increase the risk of LAS in basketball players. Dorsiflexion range of motion (DFROM) of the ankle is important in restoring reduced functional abilities and reducing the risk of re-injury. Among the talocrural antero-posterior mobilization techniques, Maitland 3rd degree talocrural anterior-posterior mobilization and Mulligan talocrural mobilization with movement are frequently preferred mobilization methods. Ankle DFROM limitation reduces the ability to absorb force through the lower extremity during jumping and landing, resulting in a decrease in vertical jumping ability. Fear of movement, called kinesiophobia, is a primary psychosocial construct in the fear-avoidance model. The development of chronic pain to sports injury appears to be a common psychological response. Because fear of re-injury can impact recovery as a barrier to return to sport, it is important to recognize fear of movement/re-injury to facilitate athletes' return to sport. Although kinesiophobia is associated with chronic orthopedic symptoms, there are no studies on athletes with LAS. There is little evidence regarding the association of kinesiophobia in athletes with chronic ankle instability, the advanced version of which presents with symptoms for 12 months or more. Although the effects of different treatment methods on kinesiophobia have been investigated in the literature, to our knowledge, the effect of talocrural joint mobilization on kinesiophobia has not been investigated. The study aimed to investigate the effects of different talocrural joint mobilization techniques on jumping performance and kinesiophobia in elite basketball players with LAS.

ELIGIBILITY:
Inclusion Criteria:

18-35 years old Being a professional basketball player Clinical diagnosis of lateral ankle sprain in the last 12 months Having a Cumberland Ankle Instability Test score <24 >2.5 cm symmetry between the two extremities in the lunge test Not to participate in any ankle treatment program in the last three months, Being Volunteer

Exclusion Criteria:

History of lower extremity surgery History of disease that may affect sensorimotor function in the lower extremity Musculoskeletal disorders that may affect balance Having any musculoskeletal and orthopedic problems Having a history of previous ankle fracture or ankle surgery Presence of any visual impairment, metabolic, neurological or rheumatological disease

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2023-07-30 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Single-leg drop jump test | baseline, immediately after the intervention
  Upon instruction, participants will aim to fall to the ground with the leg to be tested from the 30 cm high step, with their hands on their hips, and then immediately jump as high as possible. Specific instructions are given as "minimizing ground contact time and maximizing bounce height," in line with previous research. A one-minute rest is allowed between attempts.

SECONDARY OUTCOMES:
Weight-bearing lunge test | baseline, immediately after the intervention
  Weight-bearing lunge test (WBLT) is frequently used in individuals with ankle instability in order to determine dorsiflexion normal joint movement. During WBLT the participant puts their hands on the wall and takes one leg forward and the other leg helps balance behind. The maximum distance that the knee touches the wall is recorded without allowing the heel of the front foot to lose contact with the ground.
Tampa kinesiophobia scale | baseline, immediately after the intervention
  The Tampa kinesiophobia (TKS) scale is often used in musculoskeletal injuries. TKS has a checklist of 17 questions. A 4-point Likert scoring (1= I strongly disagree, 4= I totally agree) is used in the scale. After reversing items 4, 8, 12 and 16, a total score is calculated. The person gets a total score between 17-68. A high score on the scale indicates a high level of kinesiophobia.
Fear Avoidance Belief Questionnaire | baseline, immediately after the intervention
  The Fear Avoidance Questionnaire is a 10-item instrument designed to measure fear avoidance related to injury in sports. All items have a Likert type scale (1-5) from "strongly disagree" to "strongly agree" to be scored. The FAQ score ranges from 10 to 50. A higher score indicates a higher level of fear related to sports injury.

CONTACTS AND LOCATIONS:
Overall Officials: Pelin Pişirici, PT, PhD, Study Director — Bahcesehir University, Faculty of Health Sciences, Department of Physiotherapy; Arif Ozan Yıldırım, PT, MSc, Principal Investigator — Bahcesehir University, Graduate Education Institute
Locations (1):
- Bahcesehir University, Beşiktaş, Istanbul, Turkey (Türkiye)